CLINICAL TRIAL: NCT03000738
Title: The Value and Potential Mechanisms for Monocytes Subpopulations in Predicting the Prognosis of Non-Hodgkin Lymphomas.
Brief Title: The Value and Mechanisms for Monocytes Subpopulations in Predicting the Prognosis of Lymphomas
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-1163
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Lymphoma,Non-Hodgkin; Diffuse Large B Cell Lymphoma; Peripheral T-Cell Lymphoma
Keywords: CD16- monocyte/CD16+ monocyte ratio; CytoDiff flow cytometric system; Diffuse Large B Cell Lymphoma; Peripheral T-Cell Lymphoma; prognosis
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — peripheral blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- non-hodgekin lymphoma: 100 non-hodgekin lymphoma patients (age >=18y) without previous treatment would be administered, including 50 DLBCLs and 50 PTCLs.

SUMMARY:
The purpose of this study is to determine whether the CD16- monocyte/CD16+ monocyte ratio could help predict the prognosis of DLBCL and PTCL.

DETAILED DESCRIPTION:
The investigators plan to prospectively involve 100 non-hodgekin lymphoma patients, including 50 diffuse large B cell lymphomas and 50 peripheral T cell lymphomas without previous treatment from Peking Union Medical College Hospital.

The following parameters were collected: age, sex, subtype, Eastern Cooperative Oncology Group (ECOG) performance status (PS), Ann Arbor stage (I-IV), presence of B symptoms, number and type of involved sites, prognostic index including International Prognostic Index (IPI) for DLBCLand PIT for PTCL based on medical record review.

All patients would have regular treatment and follow up in PUMCH. During the follow up, treatment response was evaluated by enhanced computed tomography or PET-CT.

The peripheral blood would be collected. The Cytodiff flow cytometric technique would be used to test 16 leukocyte subpopulations from peripheral blood at the time of diagnosis, interim of treatment, end of treatment, 1 year follow-up, 1.5 year of follow-up, 2 year of follow up, 3 year of follow-up and disease progression.

Progression-free survival (PFS) and overall survival (OS) would be estimated using the Kaplan-Meier method and two-tailed log-rank test.The Cox proportional hazards model would evaluate prognostic factors for OS and PFS. Specificity, sensitivity and cut-off would be established using time-dependent receiver operating characteristic (ROC) curve analysis. Area under curve (AUC) values >0.7 indicate that the parameter can be used for diagnosis, with values >0.9 indicating high clinical accuracy.

ELIGIBILITY:
Inclusion Criteria:

1. pathologically confirmed diffuse large B cell lymphoma (DLBCL nos, PCNSL, ALK+ DLBCL, DLBCL/BL) or peripheral T cell lymphoma (AITL, ALCL, PTCL nos, NK/T nasal type, EATL, HSTL)
2. no treatment before
3. hCG(-)
4. 18 years old to 80 years old

Exclusion Criteria:

1. other tumors
2. severe infections

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed to be diffuse large B cell lymphoma or peripheral T cell lymphoma without any previous treatment in Peking Union Medical College Hospital (PUMCH) would be included.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | 3 years

SECONDARY OUTCOMES:
progression free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Daobin Zhou, MD, Study Director — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wilcox RA, Ristow K, Habermann TM, Inwards DJ, Micallef IN, Johnston PB, Colgan JP, Nowakowski GS, Ansell SM, Witzig TE, Markovic SN, Porrata L. The absolute monocyte and lymphocyte prognostic score predicts survival and identifies high-risk patients in diffuse large-B-cell lymphoma. Leukemia. 2011 Sep;25(9):1502-9. doi: 10.1038/leu.2011.112. Epub 2011 May 24. PMID 21606957
- [Background] Ziegler-Heitbrock L, Ancuta P, Crowe S, Dalod M, Grau V, Hart DN, Leenen PJ, Liu YJ, MacPherson G, Randolph GJ, Scherberich J, Schmitz J, Shortman K, Sozzani S, Strobl H, Zembala M, Austyn JM, Lutz MB. Nomenclature of monocytes and dendritic cells in blood. Blood. 2010 Oct 21;116(16):e74-80. doi: 10.1182/blood-2010-02-258558. Epub 2010 Jul 13. PMID 20628149
- [Background] Subimerb C, Pinlaor S, Lulitanond V, Khuntikeo N, Okada S, McGrath MS, Wongkham S. Circulating CD14(+) CD16(+) monocyte levels predict tissue invasive character of cholangiocarcinoma. Clin Exp Immunol. 2010 Sep;161(3):471-9. doi: 10.1111/j.1365-2249.2010.04200.x. PMID 20636398
- [Background] Heagerty PJ, Lumley T, Pepe MS. Time-dependent ROC curves for censored survival data and a diagnostic marker. Biometrics. 2000 Jun;56(2):337-44. doi: 10.1111/j.0006-341x.2000.00337.x. PMID 10877287